CLINICAL TRIAL: NCT04105920
Title: Phase III Trial Randomized to Evaluate the Interest of Hyaluronic Acid in the Preservation of Sexual Function During Prostate Curietherapies
Brief Title: Evaluation of the Interest of Hyaluronic Acid in the Preservation of Sexual Function During Prostate Curietherapies
Acronym: HYALEREC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 69HCL19_0298
Record Dates: First submitted 2019-09-10; First posted 2019-09-26 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyaluronic acid arm (Experimental): Patients included in this arm, will have, before insertion of brachytherapy seeds in the prostate, an injection of hyaluronic acid between the prostate, rectum, and pudendal arteries
  Interventions: Device: Hyaluronic acid arm
- Conventional brachytherapy (Active Comparator): Patients included in this arm will have the conventional brachytherapy.
  Interventions: Device: Hyaluronic acid arm

INTERVENTIONS:
Device: Hyaluronic acid arm — Patients included in this arm, will have, before insertion of brachytherapy seeds in the prostate, an injection of hyaluronic acid between the prostate, rectum, and pudendal arteries

SUMMARY:
Prostate cancer is the most common cancer in humans, but low mortality, around 10 / 100,000 patients / year. It differs from other cancers by its high rate of cure, as well as a long term survival. Numerous treatment techniques are available and of comparable effectiveness: as a result it must be given importance to the short and long term side effects of these different treatments.

Prostate brachytherapy with permanent implants is thus one of the standard techniques for the treatment of localized prostate cancers of favorable grades (WHO grade 1-2).

In comparison with prostatectomy and RTE, brachytherapy allows low rates of long-term urinary toxicities, and comparable rates of erectile function preservation.

With regard to erectile dysfunction, their pathophysiology after irradiation is complex and poorly understood, including damage to the erector apparatus, innervation, vascularization, and of course the level of libido.

As an example, the radiotherapy team of the Lyon Sud hospital showed that the delivering a the lowest dose of radiation to the pudendal arteries and to the penile bulb during RTE, leads to erectile preservation rates comparable with those from the literature with nearly 85% of patients with erectile function retained at 2 years . They were also able to retrospectively show that a lower dose to the pudendal arteries correlated with better erectile function during brachytherapy.

The brachytherapy procedure requires general anesthesia and endorectal ultrasound, which are optimal conditions for injecting hyaluronic acid between the prostate, rectum, and pudendal arteries. This gesture has shown to induce very few morbidity. They want to demonstrate that the injection of hyaluronic acid during prostate brachytherapy will reduce the radiation dose to the pudendal arteries and penile bulb, and thus improve the rate of preservation of erectile function in selected patients.

This randomized phase III study comparing dyserection rates after CT performed with (Arm A) and without (Arm B) injection of HA, in a patient population without erectile dysfunction before treatment.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer in humans with an incidence of about 100 / 100,000 cases / year in Europe, but low mortality, around 10 / 100,000 patients / year. It differs from other cancers by its high rate of cure, as well as a long term survival. Numerous treatment techniques are available and of comparable effectiveness: as a result it must be given importance to the short and long term side effects of these different treatments.

Prostate brachytherapy with permanent implants is thus one of the standard techniques for the treatment of localized prostate cancers of favorable grades (WHO grade 1-2). The overall survival and survival rates without biochemical recurrence at 5 and 10 years are comparable to those of other techniques such as prostatectomy or external radiotherapy (RTE), exceeding 95%.

In comparison with prostatectomy and RTE, brachytherapy allows low rates of long-term urinary toxicities, and comparable rates of erectile function preservation.

With regard to erectile dysfunction, their pathophysiology after irradiation is complex and poorly understood, including damage to the erector apparatus, innervation, vascularization, and of course the level of libido.

As an example, the radiotherapy team of the Lyon Sud hospital showed that the delivering a the lowest dose of radiation to the pudendal arteries and to the penile bulb during RTE, leads to erectile preservation rates comparable with those from the literature with nearly 85% of patients with erectile function retained at 2 years (18.5% moderate erectile dysfunction at 2 years, for moderate to severe degradation rates usually seen between 30 and 70% after external beam radiotherapy. They were also able to retrospectively show that a lower dose to the pudendal arteries correlated with better erectile function during brachytherapy.

The brachytherapy procedure requires general anesthesia and endorectal ultrasound, which are optimal conditions for injecting hyaluronic acid between the prostate, rectum, and pudendal arteries. This gesture has shown to induce very few morbidity. They want to demonstrate that the injection of hyaluronic acid during prostate brachytherapy will reduce the radiation dose to the pudendal arteries and penile bulb, and thus improve the rate of preservation of erectile function in selected patients.

This randomized phase III study comparing dyserection rates after CT performed with (Arm A) and without (Arm B) injection of HA, in a patient population without erectile dysfunction before treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years old.
* Patients over 75 years old must have a G8 score ≥ 14 or oncogeriatric assessment.The geriatrician's expertise will validate the brachytherapy treatment.
* Karnofsky performance status ≥ 60% (ECOG performance status 0-2)
* Patients diagnosed with histologically proven localized prostate adenocarcinoma
* Prostate cancer eligible for brachytherapy according to the following criteria:

  * at. Low risk prostate cancer: Gleason score <7 and PSA <10 ng / ml AND cT1-cT2a
  * Intermediate risk prostate cancers with on or two adverse factor: Gleason score = 7 (3 + 4) OR PSA 10-15ng / ml OR cT2b-cT2c / ml
  * less than 50% positive biopsies
* Volume of the prostate <60 cc
* No middle lobe
* IPSS <15/35
* Initial IIEF5 score, no treatment, greater than or equal to 20/25
* Patient able to sign an informed consent form
* Patient benefiting from a social insurance system or similar system

Exclusion Criteria:

* Nodal or distant metastatic evolution
* History of abdominal or pelvic irradiation
* Anterior treatment for prostate cancer, including hormone therapy with LHRH analogue or GnRH antagonist.
* History of prostate resection, not allowing brachytherapy seeds implantation.
* Uncontrolled cancer (except basal cell skin cancer)
* Current clinical study that may interfere with this study
* Patient unable to complete a self-administered questionnaire and understand the ins and outs of the trial
* Major patients protected by law
* Allergy to hyaluronic acid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2027-04-05 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
interest of Hyalurocnic injection to protect pudendal arteries during prostate brachytherapy in the preservation of Erectile function at 2years. | 2 years
  The primary endpoints is the comparison between the 2 groups of the proportion of patient with preserved erectile function. The erectile function will be assessed with the variation of IIEF-5 score between pre-treatment evaluation and 2years after treatment evaluation. Erectile function will be considered preserved in the absence of a decrease in the IIEF-5 score by more than 5 points.

SECONDARY OUTCOMES:
Evolution of erectile function. | 2 years
  comparison between the 2 groups of the International Index of Erectile Function (IIEF5) score evolution during the 2 years of follow-up.
The IPDE5 consumption at 2 years | 2 years
  The consumption of IPDE5 at 2 years will be defined by the proportion of patients who have used IPDE5 at least once after the intervention.
Erection satisfaction at 2 years | 2 years
  Erection satisfaction at 2 years will be measured using a numerical scale rated from 0 to 10, 0 being "not at all satisfied" and 10 "completely satisfied

OTHER OUTCOMES:
Psychosocial dimensions | 2 years
  the psychosocial dimensions of patients with erectile disfunction will be assessed using the initial EPIC (Expanded Prostate cancer Index composite / Sexual Component Questionnaire
Response assessment of IPDE5 (Phosphodiesterase 5 inhibitors ) treatement. | 6 months
  Effects Assessment of phosphodiesterase type 5 inhibitors by the EDITS (Erectile Dysfunction Inventory of Treatment Satisfaction) questionnaire 6 months after treatment.
The incidence of acute gastrointestinal and gastrourinary toxicity | 6 months
  Acute gastrointestinal and gastrointestinal toxicities are evaluated according to the V5 scale of CTCAE, initially at 6 weeks. We will evaluate the grade 2 toxicities, and the number of grade 3 or 4 toxicities in each arm.
The incidence of late gastrointestinal and gastrourinary toxicity, | 2 years
  Acute and late gastrointestinal and gastrointestinal toxicities are evaluated according to the V5 scale of CTCAE, at two years (late toxicities). We will evaluate the grade 2 toxicities, and the number of grade 3 or 4 toxicities in each arm.
Evaluation of brachytherapy by CT-MRI fusion Imaging measuring | 45 days after brachytherapy
  Quality criteria for brachytherapy will be defined on CT-MRI fusion imaging at 45 days after treatment.
Thickness hyaluronique acide injection assessment | 24 hours after surgery
  The quality of the injection of AH is defined by a thickness of AH ≥ 10 mm measured at the level of the prostatic apex.
Link between hyaluronic acid and pudendal artery stenosis. | 2 years after treatment
  The impact of hyaluronic acid injection on the probability of occurrence of pudendal artery stenosis will be assessed by centralized 2-year MRI revisions compared to MRI at day 45
Link between pudendal artheris stenosis occurrence and radiation dose received | 2 years after surgery
  The occurrence of pudendal artery stenosis (defined by centralized 2-year MRI rereading) will be correlated with the maximum dose received by these structures (Dnear max = D2% urethra, ie the minimum dose received by 2% of patients). the pudendal artery.
Link between pudendal arteries stenosis and erectile disfunction. | 2 years after treatment
  probability of occurrence of erectile dysfunction years will be correlated with the possible observation of pudendal artery stenosis at 2 years.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Jean François Leclerc, Dijon
  - Radiothérapie, Hôpital A. Michallon, CHU de Grenoble, Grenoble
  - Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No